CLINICAL TRIAL: NCT05601609
Title: Are Sporadic Colorectal Cancers in Young Distinct From Elderly?
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-2011/651-103
Record Dates: First submitted 2022-10-19; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Neoplasms
Keywords: young colorectal cancer patients; elderly colorectal cancer patients; sporadic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- young colorectal cancer (yCRC): 1. histologically confirmed cases of adenocarcinoma in the colon and rectum
  2. the age at the time of diagnosis should be ≤ 40 years
- elderly colorectal cancer (eCRC): 1. histologically confirmed cases of adenocarcinoma in the colon and rectum
  2. the age at the time of diagnosis should be ≥ 70 years

SUMMARY:
In this study, the investigators compared and evaluated the clinicopathological and oncological characteristics of sporadic colorectal cancer (CRC) in young adults without genetic mutations associated with hereditary CRC syndrome and sporadic CRC in elderly individuals.

DETAILED DESCRIPTION:
The ambiguity in the findings among several previous studies might be because of the difference in the age of the study population, yCRC and eCRC. The family history of CRC and cancer due to Crohn's disease or ulcerative colitis were also not excluded in such previous studies. Most importantly, those studies did not rule out the risk of hereditary cancer through the genetic testing in yCRC. Since hereditary CRC accounts for approximately 34% of those under the age of 35 years, it is necessary to exclude it to accurately compare the clinicopathological characteristics of sporadic cancer developed in yCRC and eCRC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cases of adenocarcinoma in the colon and rectum
* The age at the time of diagnosis should be ≤ 40 years (for yCRC) or ≥ 70 years (for eCRC)
* Genetic testing confirmation of non-hereditary cancer.

Exclusion Criteria:

* Inflammatory bowel disease
* A family history of CRC
* A history of other cancers
* Underwent any emergency operation or palliative surgery
* The Amsterdam criteria with mutations in genes associated with APC, MLH1, MSH2, MSH6

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Three tertiary referral hospitals between January 2010 to December 2017
Sampling Method: Probability Sample
Enrollment: 1599 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Overall survival outcome in young colorectal cancer (yCRC) and elderly colorectal cancer (eCRC) | The OS was defined as the time period from the date of surgery to the date of death or last follow-up up to 3 years
  The 3-year overall survival (OS) in yCRC and eCRC

SECONDARY OUTCOMES:
Cancer-specific survival outcome in young colorectal cancer (yCRC) and elderly colorectal cancer (eCRC) | CSS was defined as the time period from the date of surgery to the date of death from CRC up to 3years
  The 3-year cancer-specific survival (CSS) in yCRC and eCRC

CONTACTS AND LOCATIONS:
Overall Officials: Duck-Woo Kim, MD PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Yang IJ, Kim DW, Lee J, Ahn HM, Oh HK, Kang SB, Suh JW, Kim MH, Oh HJ, Kim HK, Kim MJ, Park JW, Ryoo SB, Park KJ, Jeong SY, Oh JH. Are sporadic colorectal cancers in young patients distinct from those in elderly patients? Colorectal Dis. 2024 Jul;26(7):1405-1414. doi: 10.1111/codi.17072. Epub 2024 Jun 16. PMID 38881232